CLINICAL TRIAL: NCT03582787
Title: Ajou University School of Medicine
Brief Title: A Comparison of McGrath MAC Videolaryngoscopy and Macintosh Laryngoscopy for Orotracheal Intubation in Children With Torticollis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-OBS-18-106
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia, Endotracheal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mcgrath group (Experimental): Orotracheal intubation with McGrath MAC videolaryngoscopy
  Interventions: Device: McGrath MAC videolaryngoscopy
- Macintosh group (Placebo Comparator): Orotracheal intubation with Macintosh laryngoscopy
  Interventions: Device: Macintosh Laryngoscopy

INTERVENTIONS:
Device: McGrath MAC videolaryngoscopy — Orotracheal intubation with McGrath MAC videolaryngoscopy after anesthetic induction
  Arms: Mcgrath group
Device: Macintosh Laryngoscopy — Orotracheal intubation with Macintosh Laryngoscopy after anesthetic induction
  Arms: Macintosh group

SUMMARY:
The primary purpose of this study is to investigate the effects of McGrath MAC videolaryngoscopy on the intubation time for orotracheal intubation in children with torticollis.

The secondary purpose of this study is to investigate the effects of McGrath MAC videolaryngoscopy on Cormack and Lehane Grade for orotracheal intubation in children with torticollis.

ELIGIBILITY:
Inclusion Criteria:

* orotracheal intubation under general anesthesia
* torticollis

Exclusion Criteria:

* •oral lesions, congenital anomaly, cervical spine instability, rapid sequence intubation

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Intubation time | through intubation completion, an average of 30 second
  Time interval between laryngoscopy passing the teeth to the confirming of end tidal CO2

SECONDARY OUTCOMES:
The degree of glottic exposure as assessed by Cormack and Lehane Grade | Up to 5 second after laryngoscopy passing the teeth
  Grade 1: full view of glottis, grade 2: Partial view of glottis, grade 3:only epiglottis seen, grade 4:neither glottis nor epiglottis seen

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Seoum, South Korea